CLINICAL TRIAL: NCT01967823
Title: Phase II Study of Metastatic Cancer That Expresses NY-ESO-1 Using Lymphodepleting Conditioning Followed by Infusion of Anti-NY ESO-1 Murine TCR-Gene Engineered Lymphocytes
Brief Title: T Cell Receptor Immunotherapy Targeting NY-ESO-1 for Patients With NY-ESO-1 Expressing Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130214; 13-C-0214
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Results first posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Melanoma; Meningioma; Breast Cancer; Non-Small Cell Lung Cancer; Hepatocellular Cancer
Keywords: Metastatic Cancer; Gene Therapy; Immunotherapy; Tumor Regression; Melanoma
MeSH Terms: conditions — Melanoma; Meningioma; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Liver Neoplasms; Neoplasm Metastasis | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/Cyclophosphamide & Fludarabine + Anti-ESO murine TCR transduced PBL + HD Aldesleukin (Experimental): Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine + anti-ESO murine T-cell receptor (TCR) transduced PBL + high-dose (HD) aldesleukin
  Interventions: Biological: Anti-NY ESO-1 mTCR PBL; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Aldesleukin

INTERVENTIONS:
Biological: Anti-NY ESO-1 mTCR PBL — Day 0: Cells will be infused intravenously (IV) on the Patient Care Unit over 20-30 minutes.
Drug: Cyclophosphamide — Days -7 and -6: Cyclophosphamide 60 mg/kg/day X 2 days intravenously (IV) in 250 mL dextrose 5% in water (D5W) infused simultaneously with mesna 15 mg/kg/day over 1 hour x 2 days.
  Other Names: Cytoxan
Drug: Fludarabine — Days -7 to -3: Fludarabine 25 mg /m^2/day intravenous piggy back (IVPB) daily over 30 minutes for 5 days.
  Other Names: Fludara
Drug: Aldesleukin — Aldesleukin 720,000 IU/kg intravenously (IV) (based on total body weight) over 15 minutes every 8 hours beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum 15 doses).
  Other Names: Proleukin

SUMMARY:
Background:

The National Cancer Institute (NCI) Surgery Branch has developed an experimental therapy for treating patients with cancer that involves taking white blood cells from the patient, growing them in the laboratory in large numbers, genetically modifying them, and then giving the cells back to the patient. In a previous study the NCI Surgery Branch used the anti-ESO-1 gene and a type of virus (retrovirus) to make these tumor fighting cells (anti-ESO-1 cells). About half of the patients who received this treatment experienced shrinking of their tumors. In this study, we are using a slightly different method of producing the anti-ESO-1 cells which we hope will be better in making the tumors shrink.

Objectives:

The purpose of this study is to see if these tumor fighting cells (genetically modified cells) that express the receptor for the ESO-1 molecule on their surface can cause tumors to shrink and to see if this treatment is safe.

Eligibility:

- Patients 15 years old and older with cancer that has the ESO-1 molecule on their tumors.

Design:

* Work up stage: Patients will be seen as an outpatient at the National Institutes of Health (NIH) clinical Center and undergo a history and physical examination, scans, x-rays, lab tests, and other tests as needed
* Leukapheresis: If the patients meet all of the requirements for the study they will undergo leukapheresis to obtain white blood cells to make the anti ESO-1 cells. {Leukapheresis is a common procedure which removes only the white blood cells from the patient.}
* Treatment: Once their cells have grown the patients will be admitted to the hospital for the conditioning chemotherapy, the anti-ESO-1 cells and aldesleukin. They will stay in the hospital for about 4 weeks for the treatment.
* Follow up: Patients will return to the clinic for a physical exam, review of side effects, lab tests, and scans about every 1-3 months for the first year, and then every 6 months to 1 year as long as their tumors are shrinking. Follow up visits take up to 2 days.

DETAILED DESCRIPTION:
PRECIS

Background:

* We have constructed a single retroviral vector that contains both and <= chains of a murine T cell receptor (mTCR) that recognizes the New York Esophageal Squamous Cell Carcinoma-1 (NY-ESO-1) (ESO) tumor antigen, which can be used to mediate genetic transfer of this T-cell receptor (TCR) with high efficiency.
* In co-cultures with human leukocyte antigen serotype within the HLA-A serotype group (HLA-A2) and ESO double positive tumors, anti-ESO mTCR transduced T cells secreted significant amounts of Interferons (IFN)- >= with high specificity.

Primary objective:

- To determine whether the administration of anti-ESO mTCR-engineered peripheral blood lymphocytes (PBL) plus high-dose aldesleukin following a non-myeloablative lymphoid depleting preparative regimen may result in objective tumor regression in patients with metastatic cancers including melanoma expressing the ESO antigen.

Eligibility:

* Age greater than or equal to 15 years and less than or equal to 70 years. Patients aged 15-17 years must weigh at least 50 kg.
* HLA-A*0201 positive
* Metastatic cancer including melanoma whose tumors express the ESO antigen
* Previously received and have been a non-responder to or recurred after receiving standard care for metastatic disease
* No contraindications for high-dose aldesleukin administration

Design:

* Peripheral blood mononuclear cells (PBMC) obtained by leukapheresis will be cultured in the presence of anti-CD3 monoclonal antibody (OKT3) and aldesleukin to stimulate T-cell growth.
* Transduction is initiated by exposure of cells to retroviral vector supernatant containing the anti-ESO mTCR genes. This mTCR targets the exact same epitope as the human T-cell receptor (hTCR).
* All patients will receive a non-myeloablative lymphocyte depleting preparative regimen of cyclophosphamide and fludarabine.
* On day 0 patients will receive anti-ESO mTCR gene-transduced PBMC and then begin high dose aldesleukin.
* A complete evaluation of evaluable lesions will be conducted 6 weeks (+/- 2 weeks) following the administration of the cell product.
* The study will be conducted using a phase II optimal design (Simon R, Controlled Clinical Trials 10:1-10, 1989). The objective will be to determine if the combination of high dose aldesleukin, lymphocyte depleting chemotherapy, and anti-ESO TCR-gene engineered lymphocytes is able to be associated with a clinical response rate that can rule out 5% (p0=0.05) in favor of a modest 20% Partial Response (PR) + Complete Response (CR) rate (p1=0.20).
* A total of up to 43 patients may be enrolled (41, plus allowing for up to 2 non-evaluable patients).

ELIGIBILITY:
* INCLUSION CRITERIA - PATIENTS WITH SOLID TUMOR CANCERS AND MELANOMA:
* Measurable (per Response Evaluation Criteria in Solid Tumors (RECIST) v1.0 criteria) metastatic cancer or locally advanced refractory/recurrent malignancy including melanoma that expresses ESO as assessed by one of the following methods: reverse transcription polymerase chain reaction (RT-PCR) on tumor tissue, immunohistochemistry of resected tissue, or serum antibody reactive with ESO.
* Confirmation of diagnosis of metastatic cancer including melanoma by the National Cancer Institute (NCI) Laboratory of Pathology.
* Patients must have previously received first-line standard therapy (or effective salvage chemotherapy regimens) for metastatic disease, if known to be effective for that disease, and have been either non-responders (progressive disease) or have recurred.
* Patients with 3 or fewer brain metastases that are less than 1 cm in diameter and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for 1 month after treatment for the patient to be eligible. Patients with surgically resected brain metastases are eligible.
* More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patient's toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).

Note: Patients may have undergone minor surgical procedures within the past three weeks, as long as all toxicities have recovered to grade 1 or less.

Note: Patients who have previously received ipilimumab and have documented gastrointestinal (GI) toxicity must have a normal colonoscopy with normal colonic biopsies.

INCLUSION CRITERIA - PATIENTS WITH MALIGNANT MENINGIOMA:

- Histologically proven recurrent meningioma or aggressive meningioma.

Note: Confirmation of ESO expression and pathology is not required in patients with definitive radiologic evidence of meningioma who are unresectable, and in whom radiation therapy without biopsy is the standard treatment.

* Recurrent disease/progression after receiving all standard treatments, which must include the following:

  * Surgical resection, if possible.
  * Definitive radiation therapy for unresectable meningioma, or for recurrent meningioma after resection.
* At least 4 weeks post-surgery, and must be at least 3 months post-radiation therapy, with resolution of related toxicities.
* Measurable disease on magnetic resonance imaging (MRI) scan.
* No history of intracranial hemorrhage.
* Patients with a history of neurofibromatosis (NF) may have other stable central nervous system (CNS) tumors, such as schwannoma, acoustic neuroma, or ependymoma only if those lesions have been stable for the past 6 months.
* Patients must be on stable dose of steroids for at least 5 days prior to baseline imaging.

INCLUSION CRITERIA - ALL PATIENTS:

* Age greater than or equal to 15 years and less than or equal to 70 years.
* Patient, or their parent(s)/legal guardian(s) (if the patient is < 18 years of age), is able to understand and willing to sign a written informed consent. Written assent will be obtained for participants under the age of 18 as appropriate.
* All participants greater than or equal to 18 years of age must be willing to sign a durable power of attorney.
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
* Patients aged 15-17 years weigh greater than or equal to 50 kg.
* Human leukocyte antigen serotype within the HLA-A serotype group (HLA-A*0201) positive.
* Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for four months after treatment.
* Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the treatment on the fetus.
* Serology

  * Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive may have decreased immune-competence and thus may be less responsive to the experimental treatment and more susceptible to its toxicities.)
  * Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be Hepatitis C Virus Ribonucleic acid(HCV RNA) negative.
* Hematology

  * Absolute neutrophil count (ANC) greater than 1000/mm(3) without the support of filgrastim
  * White blood cells (WBC) greater than or equal to 3000/mm(3)
  * Platelet count greater than or equal to 100,000/mm(3)
  * Hemoglobin greater than 8.0 g/dl. Subjects may be transfused to reach this cut-off.
* Chemistry:

  * Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than or equal to 2.5 times the upper limit of normal
  * Serum creatinine less than or equal to 1.6 mg/dl
  * Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
* Subjects must be co-enrolled in protocol 03-C-0277.

EXCLUSION CRITERIA:

* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Active systemic infections requiring anti-infective treatment, coagulation disorders, or any other active or uncompensated major medical illnesses.
* Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
* Concurrent systemic steroid therapy.
* History of severe immediate hypersensitivity reaction to cyclophosphamide, fludarabine, or aldesleukin.
* History of coronary revascularization or ischemic symptoms.
* Documented Left Ventricular Ejection Fraction (LVEF) less than or equal to 45% tested in patients:

  * Age greater than or equal to 65 years
  * With clinically significant atrial and/or ventricular arrhythmias, including but not limited to: atrial fibrillation, ventricular tachycardia, second- or third-degree heart block or have a history of ischemic heart disease and/or chest pain.
* Documented forced expiratory volume 1 (FEV1) less than or equal to 60% predicted tested in patients with:

  * A prolonged history of cigarette smoking (greater than or equal to 20 pack-year smoking history, with cessation within the past two years).
  * Symptoms of respiratory dysfunction.
* Patients who are receiving any other investigational agents.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-10-24 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenberg SA, Yang JC, Sherry RM, Kammula US, Hughes MS, Phan GQ, Citrin DE, Restifo NP, Robbins PF, Wunderlich JR, Morton KE, Laurencot CM, Steinberg SM, White DE, Dudley ME. Durable complete responses in heavily pretreated patients with metastatic melanoma using T-cell transfer immunotherapy. Clin Cancer Res. 2011 Jul 1;17(13):4550-7. doi: 10.1158/1078-0432.CCR-11-0116. Epub 2011 Apr 15. PMID 21498393
- [Background] Dudley ME, Yang JC, Sherry R, Hughes MS, Royal R, Kammula U, Robbins PF, Huang J, Citrin DE, Leitman SF, Wunderlich J, Restifo NP, Thomasian A, Downey SG, Smith FO, Klapper J, Morton K, Laurencot C, White DE, Rosenberg SA. Adoptive cell therapy for patients with metastatic melanoma: evaluation of intensive myeloablative chemoradiation preparative regimens. J Clin Oncol. 2008 Nov 10;26(32):5233-9. doi: 10.1200/JCO.2008.16.5449. Epub 2008 Sep 22. PMID 18809613
- [Background] Robbins PF, Morgan RA, Feldman SA, Yang JC, Sherry RM, Dudley ME, Wunderlich JR, Nahvi AV, Helman LJ, Mackall CL, Kammula US, Hughes MS, Restifo NP, Raffeld M, Lee CC, Levy CL, Li YF, El-Gamil M, Schwarz SL, Laurencot C, Rosenberg SA. Tumor regression in patients with metastatic synovial cell sarcoma and melanoma using genetically engineered lymphocytes reactive with NY-ESO-1. J Clin Oncol. 2011 Mar 1;29(7):917-24. doi: 10.1200/JCO.2010.32.2537. Epub 2011 Jan 31. PMID 21282551
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-C-0214.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Lymphodepleting Conditioning Foll/by Infusion of Anti-NY ESO1 Murine TCR-Gene Engineered Lymphocytes: Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine + anti-ESO murine T-cell receptor (TCR) transduced peripheral blood lymphocytes (PBL) + high-dose aldesleukin
  Anti-NY ESO-1 mTCR PBL: Day 0: Cells will be infused intravenously (IV) on the Patient Care Unit over 20-30 minutes.
  Cyclophosphamide: Days -7 and -6: Cyclophosphamide 60 mg/kg/day X 2 days intravenously (IV) in 250 mL dextrose 5% in water (D5W) infused simultaneously with mesna 15 mg/kg/day over 1 hour x 2 days.
  Fludarabine: Days -7 to -3: Fludarabine 25 mg /m^2/day intravenous piggy back (IVPB) daily over 30 minutes for 5 days.
  Aldesleukin: Aldesleukin 720,000 IU/kg intravenously (IV) (based on total body weight) over 15 minutes every 8 hours beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum 15 doses).
Period: Overall Study
Arm/Group | Lymphodepleting Conditioning Foll/by Infusion of Anti-NY ESO1 Murine TCR-Gene Engineered Lymphocytes
Started | 11
Completed | 10
Not Completed | 1
Not completed — Died prior to completing therapy (before the six-week mark). | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lymphodepleting Conditioning Foll/by Infusion of Anti-NY ESO1 Murine TCR-Gene Engineered Lymphocytes
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.43 (11.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Response
Description: Percentage of patients who have a clinical response (complete response or partial response) to treatment (objective tumor regression). Response was determined entirely by radiographic imaging using the Response Evaluation Criteria in Solid Tumors (RECIST) v1.0 to compare target lesions in centimeters. Complete Response is defined as disappearance of all target lesions. Partial Response is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD.
Time Frame: 6 and 12 weeks after cell infusion, then every 3 months x3, then every 6 months x 2, then per principal investigator (PI) discretion, up to five years or disease progression.
Population: One participant was not evaluable in terms of response.
Measure: Number; unit: percentage of participants
Arm/Group | Lymphodepleting Conditioning Foll/by Infusion of Anti-NY ESO1 Murine TCR-Gene Engineered Lymphocytes
Number analyzed (Participants) | 10
percentage of participants
  Complete Response | 10
  Partial Response | 50

2. Secondary Outcome: Percentage of T Cell Receptor (TCR) in Cluster of Differentiation 3 (CD3) + Cells
Description: T Cell Receptor (TCR) and vector presence will be quantitated in peripheral blood mononuclear cells (PBMC) samples using established polymerase chain reaction (PCR) techniques.
Time Frame: 3 and 6 months, and 1 year post cell administration
Population: Because so few patients were still on study at later time points, we felt it was more relevant to show the raw data rather than provide summary values (median, range) that could be more misleading with small numbers. Reasons participants were not analyzed: 1010004 was determined to be scientifically non-evaluable, 1010011 at 3 (± 1) mo. did not have a sample available within the time frame, and all other NA noted, were not done secondary to disease progression and/or expiration.
Measure: Number; unit: Percentage of Tcells
Groups:
- T Cell Receptor (TCR) in Cluster of Differentiation 3 (CD3) + Cells on Day of Infusion.: T Cell Receptor (TCR) in Cluster of differentiation 3 (CD3) + cells on day of infusion.
- T Cell Receptor (TCR) in Cluster of Differentiation 3 (CD3) + Cells at 3 (± 1) Months: T Cell Receptor (TCR) in Cluster of differentiation 3 (CD3) + cells at 3 (±
  1) Months
- T Cell Receptor (TCR) in Cluster of Differentiation 3 (CD3) + Cells at 6 (± 2) Months: T Cell Receptor (TCR) in Cluster of differentiation 3 (CD3) + cells at 6 (± 2) Months
- T Cell Receptor (TCR) in Cluster of Differentiation 3 (CD3) + Cells at ≥ 1 Year: T Cell Receptor (TCR) in Cluster of differentiation 3 (CD3) + cells at ≥ 1 Year
Arm/Group | T Cell Receptor (TCR) in Cluster of Differentiation 3 (CD3) + Cells on Day of Infusion. | T Cell Receptor (TCR) in Cluster of Differentiation 3 (CD3) + Cells at 3 (± 1) Months | T Cell Receptor (TCR) in Cluster of Differentiation 3 (CD3) + Cells at 6 (± 2) Months | T Cell Receptor (TCR) in Cluster of Differentiation 3 (CD3) + Cells at ≥ 1 Year
Number analyzed (Participants) | 9 | 8 | 6 | 2
Percentage of Tcells
  1010001: number analyzed (Participants) | 1 | 1 | 0 | 0
  1010001 | 81 | 1.93 |  |
  1010002: number analyzed (Participants) | 1 | 1 | 0 | 0
  1010002 | 83 | 40.9 |  |
  1010003: number analyzed (Participants) | 1 | 1 | 1 | 1
  1010003 | 76.4 | 16.1 | 7.15 | 0.87
  1010004: number analyzed (Participants) | 0 | 0 | 0 | 0
  1010005: number analyzed (Participants) | 0 | 0 | 0 | 0
  1010006: number analyzed (Participants) | 1 | 1 | 1 | 1
  1010006 | 87.3 | 16.1 | 7.15 | 0.87
  1010007: number analyzed (Participants) | 1 | 1 | 0 | 0
  1010007 | 80 | 44 |  |
  1010008: number analyzed (Participants) | 1 | 1 | 1 | 0
  1010008 | 86.7 | 16.9 | 0.28 |
  1010009: number analyzed (Participants) | 1 | 1 | 1 | 0
  1010009 | 82 | 31.8 | 18.4 |
  1010010: number analyzed (Participants) | 1 | 1 | 1 | 0
  1010010 | 68.4 | 0.37 | 0.32 |
  1010011: number analyzed (Participants) | 1 | 0 | 1 | 0
  1010011 | 78.2 |  | 46.2 |

3. Other Pre Specified Outcome: Number of Participants With Serious and Non-serious Treatment Related Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to approximately 6 weeks following cell administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Lymphodepleting Conditioning Foll/by Infusion of Anti-NY ESO1 Murine TCR-Gene Engineered Lymphocytes
Number analyzed (Participants) | 11
Participants | 11

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to approximately 6 weeks following cell administration.
Arm/Group | Lymphodepleting Conditioning Foll/by Infusion of Anti-NY ESO1 Murine TCR-Gene Engineered Lymphocytes
All-Cause Mortality (participants affected / at risk) | 8/11
Serious Adverse Events (participants affected / at risk) | 4/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lymphodepleting Conditioning Foll/by Infusion of Anti-NY ESO1 Murine TCR-Gene Engineered Lymphocytes (N=11)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (5)
Blood bilirubin increased (Blood and lymphatic system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Ejection fraction decreased (Cardiac disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Hypotension (Vascular disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 1 (1)
Urine output decreased (Renal and urinary disorders) | 1 (2)
White blood cell decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lymphodepleting Conditioning Foll/by Infusion of Anti-NY ESO1 Murine TCR-Gene Engineered Lymphocytes (N=11)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (19)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (2)
Atrial flutter (Cardiac disorders) | 1 (3)
Bilirubin (hyperbilirubinemia) (Investigations) | 3 (3)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CPK increased (Investigations) | 1 (4)
Chills (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 5 (5)
Febrile neutropenia (Investigations) | 3 (3)
Febrile neutropenia (Investigations) | 1 (1) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Fever (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Hemoglobin (Renal and urinary disorders) | 5 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (4)
Hypotension (Vascular disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (5)
INR increased (Investigations) | 1 (1)
Infection (Infections and infestations) | 2 (2) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Blood
Leukocytes (total WBC) (Investigations) | 3 (3)
Lymphocyte count decreased (Investigations) | 4 (22)
Lymphopenia (Investigations) | 7 (7)
Nausea (Gastrointestinal disorders) | 3 (6)
Neutrophil count decreased (Investigations) | 4 (10)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 7 (7)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (1)
Platelet count decreased (Investigations) | 4 (12)
Platelets (Investigations) | 7 (7)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Restlessness (Nervous system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Urine output decreased (Renal and urinary disorders) | 2 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (3)
Weight loss (Investigations) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 4 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT01967823/Prot_SAP_000.pdf
  • Informed Consent Form: Standard (2018-08-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT01967823/ICF_001.pdf
  • Informed Consent Form: Assent (2018-08-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT01967823/ICF_002.pdf